CLINICAL TRIAL: NCT01732926
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Idelalisib (GS-1101) in Combination With Bendamustine and Rituximab for Previously Treated Indolent Non-Hodgkin Lymphomas
Brief Title: Efficacy and Safety of Idelalisib (GS-1101) in Combination With Bendamustine and Rituximab for Previously Treated Indolent Non-Hodgkin Lymphomas
Acronym: Bridalveil
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-313-0125; 2012-004034-42 (EudraCT Number)
Record Dates: First submitted 2012-11-14; First posted 2012-11-26 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2017-03

CONDITIONS: Indolent Non-Hodgkin's Lymphomas
Keywords: iNHL; indolent NHL; follicular lymphoma; CAL-101; rituximab; bendamustine; small lymphocytic lymphoma; lymphoplasmacytoid lymphoma; Waldenstrom macroglobulinemia; LPL; WM; Marginal zone lymphoma; MZL; SLL; FL; GS-1101; PI3K inhibitor; idelalisib
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone | interventions — idelalisib; Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rituximab + Bendamustine + Idelalisib (Experimental): Participants will receive rituximab + bendamustine + idelalisib.
  Interventions: Drug: Idelalisib; Drug: Rituximab; Drug: Bendamustine
- Rituximab + Bendamustine + Placebo (Experimental): Participants will receive rituximab + bendamustine + placebo.
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Placebo

INTERVENTIONS:
Drug: Idelalisib — 150 mg tablet administered orally twice daily
  Other Names: Zydelig®; CAL-101; GS-1101
  Arms: Rituximab + Bendamustine + Idelalisib
Drug: Rituximab — 375 mg/m^2 single-use vials administered intravenously every 4 weeks (up to a total of 6 infusions)
  Other Names: Rituxan®; MabThera®
Drug: Bendamustine — 90 mg/m^2 single-use vials administered intravenously for two consecutive days every 4 weeks (up to a total of 4-6 cycles as tolerated)
  Other Names: Treanda®
Drug: Placebo — Tablet administered orally twice daily
  Arms: Rituximab + Bendamustine + Placebo

SUMMARY:
The primary objective of this study is to evaluate the addition of idelalisib to bendamustine/rituximab on progression-free survival (PFS) in adults with previously treated indolent non-Hodgkin lymphoma (iNHL).

An increased rate of deaths and serious adverse events (SAEs) among participants with front-line chronic lymphocytic leukemia (CLL) and early-line iNHL treated with idelalisib in combination with standard therapies was observed by the independent data monitoring committee (DMC) during regular review of 3 Gilead Phase 3 studies. Gilead reviewed the unblinded data and terminated this study in agreement with the DMC recommendation and in consultation with the US Food and Drug Administration (FDA).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of B-cell iNHL, with histological subtype limited to the following

  1. Follicular lymphoma (FL) Grade 1, 2, or 3a
  2. Small lymphocytic lymphoma (SLL)
  3. Lymphoplasmacytoid lymphoma/Waldenström macroglobulinemia (LPL/WM)
  4. Marginal zone lymphoma (MZL) (splenic, nodal, or extra-nodal)

Key Exclusion Criteria:

* History of lymphoid malignancy other than those allowed per inclusion criteria.
* Ongoing drug-induced liver injury, active hepatitis C, active hepatitis B, alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, or portal hypertension.
* Prior treatment with bendamustine that was not effective.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2013-01-02 (Actual); Primary Completion 2016-05-17 (Actual); Study Completion 2016-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (144):
- United States (33):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - Comprehensive Blood and Cancer Center (Bakersfield), Bakersfield, California
  - Saint Jude Heritage Healthcare (TORI), Fullerton, California
  - Pacific Shores Medical Group, Long Beach, California
  - Cancer Care Associates, Redondo Beach, California
  - San Luis Obispo Oncology and Hematology, San Luis Obispo, California
  - Cancer Center of Santa Barbara, Santa Barbara, California
  - Central Coast Medical Oncology Group, Santa Maria, California
  - St Joseph Heritage Healthcare System, Santa Rosa, California
  - Kaiser Permanente Vallejo Medical Center, Vallejo, California
  - Sylvester Comprehensive Cancer Center/UMHC, Deerfield Beach, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Joliet Oncology Hematology Associates Ltd., Joliet, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - North Shore Hematology/Oncology Associates, East Setauket, New York
  - Weill Cornell Medical College, New York, New York
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Hollings Cancer Center, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Greenville, South Carolina
  - Texas Oncology, P.A., Bedford, Texas
  - Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology, P.A., Denton, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Texas Oncology, P.A., Harlingen, Texas
  - Texas Oncology, P.A., Weslaco, Texas
  - Swedish Medical Center, Seattle, Washington
  - Northwest Medical Specialists, Tacoma, Washington
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (9):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Haematology and Oncology Clinics of Australia Gold Coast, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Saint Vincent's Hospital, Fitzroy, Victoria
  - Western Hospital, Footscray, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Canada (12):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Fraser Clinical Trials, Inc., New Westminster, British Columbia
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Centre for Clinical Research, Halifax, Nova Scotia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hôpital Charles Lemoyne, Greenfield Park, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre Hospitalier Affilie Universitaire de Quebec, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - CancerCare Manitoba, Winnipeg
- Czechia (3):
  - Fakultní Nemocnice Ostrava, Ostrava - Poruba, Severomoravsky KRAJ
  - Fakultní nemocnice Brno, Brno
  - Fakultní nemocnice Hradec Králové, Hradec Králové
- France (16):
  - CHR Metz, Metz, Alsace
  - Centre Hospitalier Universitaire de Strasbourg - Hôpital Hautepierre, Strasbourg, Alsace
  - Institut Bergonié, Bordeaux, Aquitaine
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Centre Henri-Becquerel, Rouen, Haute-normandie
  - Centre Jean Bernard, Le Mans, Pays de la Loire Region
  - Centre Hospitalier Universitaire Brest, Brest
  - Centre Hospitalier de Dunkerque, Dunkirk
  - Centre Hospitalier Départmental La Roche sur Yon, La Roche-sur-Yon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital Hôtel-Dieu, Nantes
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Régional et Universitaire - Hôpital Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif
  - Hôpital Necker-Enfants Malades, Paris, Île-de-France Region
- Germany (5):
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen, Baden-Wurttemberg
  - Gemeinschaftspraxis Dres. Söling Und Siehl, Kassel, Hesse
  - Vivantes Klinikum am Urban, Berlin
  - Charite - Campus Virchow, Berlin
  - Klinikum der Ludwig-Maximilians-Universität München, München
- Israel (4):
  - Barzilai Medical Center, Ashkelon
  - Soroka University Medical Center, Beersheba
  - Rambam Health Corp., Haifa
  - Hadassah Medical Organization, Ein Kerem, Jerusalem
- Italy (11):
  - Centro di Riferimento Oncologico di Aviano, Aviano
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Spedali Civili Di Brescia Azienda Ospedaliera, Brescia
  - IRCCS Azienda Ospedaliera Universitaria San Martino, Genova
  - Ospedale San Raffaele-IRCCS, Milan
  - Azienda Ospedaliera Ospedale Niguarda Ca' Granda, Milan
  - Azienda Ospedaliero Universitaria (AOU) "Maggiore della Carita" di Novara, Novara
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro
  - Azienda Unità Sanitaria Locale di Piacenza-Ospedale Guglielmo da Saliceto, Piacenza
  - Azienda Ospedaliera Universitaria Senese - Policlinico S. Maria alle Scotte, Siena
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Poland (9):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Malopolskie Centrum Medyczne S.C., Krakow
  - Wojewódzki Szpital Specjalistyczny im. Mikolaja Kopernika w Lodzi, Lódz
  - Szpital Kliniczny nr 1, Katedra i Klinika Hematoonkologii i Transplantacji Szpiku, Lublin
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Ministerstwa Spraw Wewnetrznych z Warminsko-Mazurskim, Olsztyn
  - Wojewódzki Szpital Specjalistyczny im. Janusza Korczaka w Slupsku, Słupsk
  - Centralny Szpital Kliniczny MSW w Warszawie, Warsaw
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Centrum Onkologii i Hipertermii, Warsaw
- Russia (10):
  - N. N. Blokhin Russian Cancer Research Center, Moscow
  - Nizhny Novgorod Regional Clinical Hospital n.a. N.A. Semashko, Nizhny Novgorod
  - Ryazan Regional Clinical Hospital, Ryazan
  - FGU Russian Scientific Research Institute of Hematology and Transfusiology, Saint Petersburg
  - Saint Petersburg I.P. Pavlov State Medical University, Saint Petersburg
  - FSI "V.A. Almazov Federal Centre of Heart, Blood and Endocrinology of Rosmedtechnologies", Saint Petersburg
  - Saratov State Medical University, Saratov
  - State Budgetary Healthcare Institution "Volgograd Regional Clinical Oncology Dispensary #1", Volgograd
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
  - Central City Hospital # 7, Yekaterinburg
- South Korea (4):
  - Dong-A University Medical Center, Busan
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (8):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitario La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fé de Valencia, Valencia
- Sweden (2):
  - Karolinska Universitetssjukhuset, Huddinge, Stockholm County
  - Länssjukhuset Ryhov, Jönköping
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - China Medical University Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (14):
  - Kent and Canterbury Hospital, Canterbury, England
  - University Hospital Coventry, Coventry, England
  - Royal Bournemouth General Hospital, Dorset, England
  - Leeds Teaching Hospitals NHS Trust, Leeds, England
  - Barts and The London NHS Trust, London, England
  - University College London Hospitals National Health Society Foundation Trust, London, England
  - Guys and Saint Thomas NHS Foundation Trust, London, England
  - Imperial College Healthcare NHS Trust, London, England
  - Maidstone Hospital, Maidstone, England
  - Christie Hospital NHS Foundation Trust, Manchester, England
  - Oxford University Hospitals NHS Trust, Oxford, England
  - Southampton General Hospital, Southampton, England
  - Mount Vernon Hospital, Middlesex
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the North America, Europe, and Asia Pacific. The first participant was screened on 02 January 2013. The last study visit occurred on 17 May 2016.
Pre-assignment Details: 581 participants were screened.
Groups:
- Idelalisib + Bendamustine + Rituximab: Idelalisib (Zydelig®) 150 mg tablet twice daily + bendamustine intravenously (starting dose of 90 mg/m^2 for up to 12 infusions)
  + rituximab intravenously (375 mg/m^2 on Day 1 for a total of 6 infusions)
- Placebo + Bendamustine + Rituximab: Placebo tablet twice daily + bendamustine intravenously (starting dose of 90 mg/m^2 for up to 12 infusions) + rituximab intravenously (375 mg/m^2 on Day 1 for a total of 6 infusions)
Period: Overall Study
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab
Started | 320 | 155
Completed (Completed = reached primary efficacy endpoint of progressive disease or death) | 53 | 45
Not Completed | 267 | 110
Not completed — Study Terminated by Sponsor | 168 | 80
Not completed — Withdrawal by Subject | 46 | 8
Not completed — Physician Decision | 24 | 11
Not completed — Other Reason | 21 | 4
Not completed — Initiation of Other Anti-Cancer Therapy | 7 | 6
Not completed — Blind Broken by Subject or Study Site | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) Analysis Set: all participants who were randomized regardless of whether they received any study treatment
Groups:
- Idelalisib + Bendamustine + Rituximab: Idelalisib 150 mg tablet twice daily + bendamustine intravenously (starting dose of 90 mg/m^2 for up to 12 infusions) + rituximab intravenously (375 mg/m^2 on Day 1 for a total of 6 infusions)
- Total: Total of all reporting groups
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab | Total
Number analyzed (Participants) | 320 | 155 | 475
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (10.5) | 62 (11.1) | 62 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 58 | 190
  Male | 188 | 97 | 285
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 26 | 8 | 34
  Black or African American | 2 | 2 | 4
  White | 247 | 122 | 369
  Other | 4 | 2 | 6
  Not Permitted | 41 | 21 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 8 | 24
  Not Hispanic or Latino | 262 | 129 | 391
  Not Permitted | 42 | 18 | 60
Region of Enrollment [Count of Participants; unit: Participants]
  Russian Federation | 16 | 11 | 27
  United States | 37 | 12 | 49
  United Kingdom | 33 | 20 | 53
  Spain | 21 | 11 | 32
  Canada | 47 | 19 | 66
  Czech Republic | 12 | 7 | 19
  Sweden | 3 | 2 | 5
  Taiwan | 7 | 2 | 9
  Poland | 25 | 11 | 36
  Korea, Republic of | 10 | 2 | 12
  Italy | 21 | 14 | 35
  Israel | 6 | 2 | 8
  France | 36 | 18 | 54
  Australia | 44 | 23 | 67
  Germany | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the interval from randomization to the earlier of the first documentation of definitive indolent non-Hodgkin lymphomas (iNHL) disease progression or death from any cause. Definitive iNHL disease progression is progression based on standard criteria. PFS was to be assessed by an independent review committee (IRC).
Population: Due to the early termination of the study, efficacy data were not available for all participants, and therefore the prespecified analyses were not conducted.
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Complete Response Rate (CR)
Description: Complete response rate is defined as the proportion of participants who achieve a complete response. CR rate was to be assessed by an IRC.
Population: as for outcome 1
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate is defined as the proportion of participants who achieve a complete response or partial response (or very good partial response (VGPR) or minor response (MR) for participants with Waldenstrom's). ORR was to be assessed by an IRC.
Population: as for outcome 1
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Lymph Node Response Rate
Description: Lymph node response rate is defined as the proportion of participants who achieve ≥ 50% decrease from baseline in the sum of the products of the greatest perpendicular diameters of index lesions. Lymph node response rate was to be assessed by an IRC.
Population: as for outcome 1
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the interval from randomization to death from any cause.
Population: Due to the early termination of the study, efficacy data were not mature for all participants, and therefore the prespecified analyses were not conducted.
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 34 months plus 30 days
Description: Safety Analysis Set: all participants who took at least 1 dose of study drug
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab
Serious Adverse Events (participants affected / at risk) | 229/317 | 58/155
Other Adverse Events (participants affected / at risk) | 315/317 | 147/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib + Bendamustine + Rituximab (N=317) | Placebo + Bendamustine + Rituximab (N=155)
Anaemia (Blood and lymphatic system disorders) | 8 | 4
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 45 | 7
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 8 | 3
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Dilatation ventricular (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Ophthalmoplegia (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Colitis (Gastrointestinal disorders) | 9 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 14 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Chills (General disorders) | 2 | 0
Death (General disorders) | 1 | 0
Device related thrombosis (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Hypothermia (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 2
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 67 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 2 | 0
Hepatocellular injury (Hepatobiliary disorders) | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 3 | 1
Hypersensitivity (Immune system disorders) | 4 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Campylobacter infection (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 5 | 1
Clostridium difficile colitis (Infections and infestations) | 3 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 2 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Cytomegalovirus hepatitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 6 | 0
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 0 | 1
Enteritis infectious (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 2
Gingivitis (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 2 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Infectious colitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 4 | 1
Listeria sepsis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 5 | 3
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 3 | 0
Neutropenic sepsis (Infections and infestations) | 4 | 2
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Otitis media chronic (Infections and infestations) | 1 | 1
Pneumocystis jirovecii infection (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 9 | 0
Pneumonia (Infections and infestations) | 24 | 4
Pneumonia bacterial (Infections and infestations) | 2 | 0
Pneumonia chlamydial (Infections and infestations) | 1 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2
Salmonellosis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 9 | 1
Septic shock (Infections and infestations) | 2 | 2
Sinusitis (Infections and infestations) | 3 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Systemic mycosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 0
Urinary tract infection (Infections and infestations) | 6 | 1
Urosepsis (Infections and infestations) | 2 | 0
Varicella (Infections and infestations) | 3 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 3
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Sacroiliac fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 14 | 0
Aspartate aminotransferase increased (Investigations) | 12 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 3
Transaminases increased (Investigations) | 2 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Richter's syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Complex regional pain syndrome (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Mixed dementia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 6 | 2
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 16 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 18 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1
Embolism (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
Internal haemorrhage (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib + Bendamustine + Rituximab (N=317) | Placebo + Bendamustine + Rituximab (N=155)
Anaemia (Blood and lymphatic system disorders) | 51 | 18
Leukopenia (Blood and lymphatic system disorders) | 18 | 7
Neutropenia (Blood and lymphatic system disorders) | 122 | 54
Thrombocytopenia (Blood and lymphatic system disorders) | 37 | 18
Abdominal pain (Gastrointestinal disorders) | 39 | 11
Abdominal pain upper (Gastrointestinal disorders) | 21 | 10
Constipation (Gastrointestinal disorders) | 74 | 31
Diarrhoea (Gastrointestinal disorders) | 158 | 33
Dry mouth (Gastrointestinal disorders) | 20 | 3
Dyspepsia (Gastrointestinal disorders) | 28 | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 17 | 6
Mouth ulceration (Gastrointestinal disorders) | 20 | 4
Nausea (Gastrointestinal disorders) | 159 | 65
Stomatitis (Gastrointestinal disorders) | 26 | 5
Vomiting (Gastrointestinal disorders) | 100 | 25
Asthenia (General disorders) | 43 | 24
Chills (General disorders) | 39 | 10
Fatigue (General disorders) | 103 | 51
Mucosal inflammation (General disorders) | 29 | 2
Oedema peripheral (General disorders) | 38 | 7
Pyrexia (General disorders) | 135 | 22
Bronchitis (Infections and infestations) | 22 | 13
Herpes zoster (Infections and infestations) | 19 | 7
Lower respiratory tract infection (Infections and infestations) | 14 | 9
Nasopharyngitis (Infections and infestations) | 17 | 14
Oral candidiasis (Infections and infestations) | 17 | 2
Pneumonia (Infections and infestations) | 16 | 2
Sinusitis (Infections and infestations) | 18 | 11
Upper respiratory tract infection (Infections and infestations) | 58 | 25
Urinary tract infection (Infections and infestations) | 26 | 8
Infusion related reaction (Injury, poisoning and procedural complications) | 38 | 16
Alanine aminotransferase increased (Investigations) | 65 | 3
Aspartate aminotransferase increased (Investigations) | 51 | 4
Neutrophil count decreased (Investigations) | 12 | 9
Weight decreased (Investigations) | 41 | 6
Decreased appetite (Metabolism and nutrition disorders) | 65 | 25
Hypokalaemia (Metabolism and nutrition disorders) | 52 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 19 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 8
Dizziness (Nervous system disorders) | 23 | 10
Dysgeusia (Nervous system disorders) | 16 | 10
Headache (Nervous system disorders) | 45 | 18
Neuropathy peripheral (Nervous system disorders) | 8 | 9
Paraesthesia (Nervous system disorders) | 9 | 9
Insomnia (Psychiatric disorders) | 40 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 71 | 37
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 20 | 5
Erythema (Skin and subcutaneous tissue disorders) | 20 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 16 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 54 | 22
Rash (Skin and subcutaneous tissue disorders) | 105 | 16
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 29 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 16 | 4
Hypotension (Vascular disorders) | 16 | 5

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, efficacy data were not available for all participants, and therefore the prespecified analyses were not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years